CLINICAL TRIAL: NCT03986567
Title: Impact of New Communication Technologies and Gamification in the Promotion of Partner Notification of Sexually Transmitted Infections Among Young People: The "Notijoves" Randomised Controlled
Brief Title: The "Notijoves" Randomised Controlled
Acronym: notijoves
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 40547236
Record Dates: First submitted 2018-11-15; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2018-10

CONDITIONS: Sexually Transmitted Diseases
Keywords: Mobile Applications; Contact Tracing; Game Theory; Adolescent
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Active Comparator): Providing with a paper notification card to the STI diagnosed young person
  Interventions: Behavioral: gamification for partner notification among youngsters
- intervention web app (Experimental): providing to the STI diagnosed young person, with a code number to enter into the app to notify sexual partners
  Interventions: Behavioral: gamification for partner notification among youngsters
- intervention game (Experimental): providing to the STI diagnosed young person, with a code number to enter into the app and play a game to get motivated to notify sexual partners
  Interventions: Behavioral: gamification for partner notification among youngsters

INTERVENTIONS:
Behavioral: gamification for partner notification among youngsters — Design a web based tool adapted to Mobile phones for partner notification of STI among youngsters 16 to 24 years old and evaluate its role in increasing the "patient referral" partner notification

SUMMARY:
Background:

Increase of sexually transmitted infections (STIs) as well as increased use of new information and communication technologies (ICTs) among young people in Catalonia triggers the idea of designing a mobile phone application to promote partner notification.

Objective:

Design a web based tool adapted to Mobile phones for partner notification of STI among youngsters 16 to 24 years old and evaluate its role in increasing the "patient referral" partner notification.

Methods:

This is a multicentre randomised controlled trial with a proportional stratification of the sample by centre and random allocation of participants to the three arms of the study (simple web based intervention, game web based intervention and control). This study is conducted by midwives, gynaecologists and physicians in the sexual and reproductive areas of the primary health care centres.

The study population is: 1- All youngsters 16 to 24 years old diagnosed with one of the three curable STIs, (Syphilis, gonococcus and chlamydia). 2- All partners of those diagnosed with the previous STIs, independently of their state of infection.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 24 years old diagnosed with one of the three curable STIs, (Syphilis, gonococcus and chlamydia).
* All partners of those diagnosed with the previous STIs, independently of their state of infection.

Exclusion Criteria:

* Already participated in the study within its length

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 416 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of partner notification: number of partners notified out of number of cases diagnosed | 2 months after diagnose
  number of partners notified out of number of cases diagnosed

SECONDARY OUTCOMES:
yield of early diagnosis and treatment of those exposed and infected; | 3 months
  number of partners exposed out of number of cases diagnosed

CONTACTS AND LOCATIONS:
Overall Officials: GEMMA FALGUERA PUIG, PhD, Principal Investigator — CATALAN INSTITUTE OF HEALTH (ICS)
Locations (1):
- Catalan Institute of Health (Ics), Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No